CLINICAL TRIAL: NCT04803773
Title: MRI-guided Focused Ultrasound for Bone Tumors Treatment: Feasibility Study for the Treatment of Bone Metastases and osteoïd Osteoma
Brief Title: MRI-guided Focused Ultrasound : Feasibility Study for the Treatment of Bone Metastases and osteoïd Osteoma
Acronym: UFOGUIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 7677
Record Dates: First submitted 2021-01-05; First posted 2021-03-18 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Painful Bone Metastases; Superficial Osteoid Osteoma
Keywords: thermal ablation; HIFU; Bone metastases; Osteoid Osteoma; Pain; Interventional Radiology
MeSH Terms: conditions — Osteoma, Osteoid; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Device: UFOGUIDE "patient transducer"

INTERVENTIONS:
Device: UFOGUIDE "patient transducer" — The transducer is maintained by a flexible/rigid structure, consisting of a support base, and three to four feet forming an arch around the area to be treated. These feet exist in several lengths (10, 20, 30, 40 cm) depending on the area to be treated and can be easily mounted on the base by fast attachment. The structure is based on the principle of granular jamming: it is flexible in its normal state, and can be stiffened by the application of depression within the feet.

SUMMARY:
Ufoguide is a prospective single arm open study to assess the feasibility of a new type of HIFU system to treat bone tumors.

HIFU is classically delivered by a transducer integrated in the MRI table. This study assesses a new type of approach in which the HIFU transducer is manually placed on the skin of the patient, under the assistance of optical navigation, and held in place by MR-compatible passive arms.

The primary goal of this study is to assess the feasibility of heating the tumor accurately with this new HIFU system. The evaluation and monitoring of the treatment will be performed by MR thermometry.

Secondary endpoints include the evaluation of clinical efficacy, quality of life and safety.

DETAILED DESCRIPTION:
Ufoguide is a prospective single arm open study to assess the feasibility of a new type of HIFU system for the treatment of painful metastases (palliative intent) and osteoid osteoma (curative intent).

HIFU is classically delivered by a transducer integrated in the MRI table. This study assesses a new type of approach in which the HIFU transducer is manually placed on the skin of the patient and held in place by MR-compatible passive arms. Optical infrared navigation is used to help the physician with the positioning of the HIFU transducer.

The primary goal of this study is to assess the feasibility of heating the tumor accurately with this new HIFU system. The evaluation and control of the treatment will be performed by Proton Resonance Frequency Shift (PRFS) MR thermometry.

Secondary endpoints include the evaluation of clinical efficacy, quality of life and safety.

Clinical efficacy is defined:

* in palliative intent by a decrease ≤3 on visual analogic scale
* in curative intent (osteoid osteoma) by a total disappearance of pain Quality of life is assessed by EORTC quality of life questionnaire-core 30 items Complications are recorded to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject with one or more painful bone metastases (EVA≥5)
* Subject with sub-perolate or cortical osteoid osteoma
* For people with painful bone metastases: first-line treatment or radiotherapy failure
* Weight < 140kg.
* Target tumor accessible by HIFU-MRI
* Maximum size of the lesion - 20cm²
* Depth of the lesion to be treated - 4mm and 10cm
* Subject affiliated with a health insurance social protection.
* A subject capable of understanding research objectives and risks and giving informed and signed consent
* Subject who has been informed of the pre-medical visit results

Exclusion Criteria:

* MRI contraindication
* Contraindication to the use of a gadolinium contrast or hypersensitivity to gadoteric acid, meglumine or any drug containing gadolinium
* General anesthesia contraindication
* Non-reversible hemostasis disorders
* Previous injury on the area to be treated (radiotherapy, surgery, ...)
* Tumors located on the spine or skull
* Tumors located on the ribs
* Pathological fracture
* For Osteoid Osteoma: nidus more than 1cm deep within cortical bone
* Pregnant woman (pregnancy test, urinary or HCG dosage, negative to inclusion) or lactating
* existence of dermatological pathologies
* Subject with a known latex allergy
* Subject under safeguarding of justice, under guardianship or curatorship
* Subject in an exclusion period by a previous or ongoing study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-11-09 (Estimated); Study Completion 2024-11-09 (Estimated)

PRIMARY OUTCOMES:
Device feasibility | Assessed in real time during the procedure
  The device feasibility is defined by the ability of the device to induce a hyperthermia on the tumor

SECONDARY OUTCOMES:
Clinical efficacy: - in palliative intent by a decrease ≤3 on visual analogic scale - in curative intent (osteoid osteoma) by a total disappearance in pain | Before intervention and day 1, day 5 and day 30
  Clinical efficacy is defined:
  * in palliative intent by a decrease ≤3 on visual analogic scale
  * in curative intent (osteoid osteoma) by a total disappearance in pain
Quality of life using the EORTC (European Organisation for Research and Treatment of Cancer) quality of life questionnaire | Before intervention and day 30
  EORTC quality of life questionnaire is composed of multi-items scales and single-item measures. All of the scales measures range in score from 0 to 100. A High scale score represents a higher response level.
Safety :number of patients with complications and characterization of complications | day 1, day 5 and day 30
  Complications recording

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No